CLINICAL TRIAL: NCT01715896
Title: A Phase 2 Exploratory Study of Mavrilimumab Versus Anti-tumor Necrosis Factor in Subjects With Rheumatoid Arthritis
Brief Title: A Study of Mavrilimumab Versus Anti Tumor Necrosis Factor in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-IA-CAM-3001-1107
Record Dates: First submitted 2012-10-16; First posted 2012-10-29 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Golimumab; Mavrilimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — golimumab; mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Golimumab 50 mg alternating with Placebo (Experimental): Participants received alternating doses of golimumab 50 milligram (mg) (Weeks 0, 4, 8, 12, 16, 20, and 24) and placebo matched to mavrilimumab (Weeks 2, 6, 10, 14, 18, and 22) injections subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Interventions: Biological: Golimumab 50 mg
- Mavrilimumab 100 mg (Experimental): Participants received Mavrilimumab 100 mg injection subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Interventions: Biological: Mavrilimumab 100 mg

INTERVENTIONS:
Biological: Golimumab 50 mg — Participants received alternating doses of golimumab 50 mg (Weeks 0, 4, 8, 12, 16, 20, and 24) and placebo matched to mavrilimumab (Weeks 2, 6, 10, 14, 18, and 22) injections subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Arms: Golimumab 50 mg alternating with Placebo
Biological: Mavrilimumab 100 mg — Participants received Mavrilimumab 100 mg injection subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
  Other Names: CAM-3001
  Arms: Mavrilimumab 100 mg

SUMMARY:
The primary objectives of this study is to explore the efficacy of mavrilimumab compared with golimumab in the treatment of adult subjects 18-80 years of age with moderate-to-severe active rheumatoid arthritis (RA) who have an inadequate response to one or more conventional disease-modifying anti-rheumatic drugs (DMARDs) and/or one or two anti-tumor necrosis factor (TNF) agents (excluding golimumab) for efficacy or safety reasons.

DETAILED DESCRIPTION:
Despite the therapeutic improvements with recent biologic agents approved for rheumatoid arthritis (RA), there is still a significant unmet medical need for the treatment of subjects with this chronic disease to achieve a faster, more complete response, and higher rates of remission. The aim of the current study is to compare the efficacy and safety of a subcutaneous dose of mavrilimumab with a marketed treatment for RA (golimumab) in 120 adult subjects with moderate-to-severe active RA who have had an inadequate response to one or two anti-TNF agents with mavrilimumab. The design of the study was exploratory and not formerly statistically powered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 80 years
* Written consent
* Diagnosis of adult onset Rheumatoid Arthritis (RA) as defined by the 2010 American College of Rheumatology European League Against Rheumatism (ACR/EULAR) classification criteria
* Moderately active disease as defined by disease activity score in 28 joints C-reactive protein (DAS28[CRP]) greater than or equal to (>=) 3.2 at screening and DAS28 erythrocyte sedimentation rate(ESR) ≥ 3.2 at Day 1
* Inadequate response to one or more conventional disease-modifying anti-rheumatic drugs (DMARDs)
* At least 4 swollen joints
* Inadequate response to one or two anti-TNF agents other than the study comparator, as defined by the protocol
* Receiving oral or injectable methotrexate, as defined by the protocol.

Exclusion Criteria:

* A rheumatic autoimmune disease or other inflammatory joint disease other than RA
* Previous treatment with biologic therapies other than anti-TNF for RA
* Treatment with other DMARDs or non-steroidal anti-inflammatory drugs (NSAIDs), as defined by the protocol.
* Medical history as defined by the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Albulescu, Study Director — MedImmune Ltd
Locations (39):
- Argentina (3):
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Córdoba
  - Research Site, San Miguel de Tucumán
- Research Site, Barranquilla, Colombia
- Czechia (3):
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Research Site, Montpellier, France
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Larissa
- Hungary (3):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Rehovot
- Research Site, Mérida, Mexico
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Viseu
- Russia (3):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niška Banja
- Slovakia (3):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Kosice - Saca
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Málaga
- United Kingdom (5):
  - Research Site, Birkenhead
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Plymouth

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 215 participants were screened, of which 77 participants were considered as screen failures and 138 participants were randomized and completed in the study.
Groups:
- Golimumab 50 Milligram (mg) Alternating With Placebo: Participants received alternating doses of golimumab 50 mg (Weeks 0, 4, 8, 12, 16, 20, and 24) and placebo matched to mavrilimumab (Weeks 2, 6, 10, 14, 18, and 22) injections subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
Period: Overall Study
Arm/Group | Golimumab 50 Milligram (mg) Alternating With Placebo | Mavrilimumab 100 mg
Started | 68 | 70
Completed | 65 | 59
Not Completed | 3 | 11
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Population: The modified intent to treat (mITT) population analysis set included all participants in the treatment group corresponding to their randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Golimumab 50 Milligram (mg) Alternating With Placebo | Mavrilimumab 100 mg | Total
Number analyzed (Participants) | 68 | 70 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.4) | 50.2 (13.3) | 50.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 113
  Male | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 20 (ACR20) Responses at Day 169
Description: The ACR20 was defined as greater than or equal to (>=) 20 percent (%) improvement, in: swollen joint count (SJC) and tender joint count (TJC) and >=20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity (PGA); physician global assessment of disease activity (MDGA); self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-reactive protein (CRP). If CRP was missing and Erythrocyte sedimentation rate (ESR) was present then ESR was to be used.
Time Frame: Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group.
Measure: Number; unit: percentage of participants
Groups:
- Golimumab 50 mg Alternating With Placebo: Participants received alternating doses of golimumab 50 mg (Weeks 0, 4, 8, 12, 16, 20, and 24) and placebo matched to mavrilimumab (Weeks 2, 6, 10, 14, 18, and 22) injections subcutaneously every 2 weeks for 24 weeks in combination with stable dose of methotrexate (7.5 to 25 mg per week) through oral or parenteral route.
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 65.6 | 62.0
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.666, Logit response Model; Percent difference = -3.5, 90% CI 2-sided [-16.8 to 9.8] — P-value and 90% unconditional exact confidence interval (CI) was calculated using the model of logit (response) = strata + treatment

2. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 50 (ACR50) Responses at Day 169
Description: The ACR50 was defined as >=50% improvement, in: SJC and TJC and >=50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP. If CRP was missing and ESR was present then ESR was to be used. The percentage of participants were calculated by logistic regression model method.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 43.4 | 34.8
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.293, Logit response Model; Percent difference = -8.6, 90% CI 2-sided [-22.0 to 4.8] — P-value and 90% unconditional exact CI was calculated using the model of logit (response) = strata + treatment

3. Primary Outcome: Percentage of Participants Who Achieved American College of Rheumatology 70 (ACR70) Responses at Day 169
Description: The ACR70 was defined as >=70% improvement, in: SJC and TJC and >=70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP. If CRP was missing and ESR was present then ESR was to be used. The percentage of participants were calculated by logistic regression model method.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 25.9 | 16.1
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.156, Logit Response Model; Percent difference = -9.8, 90% CI 2-sided [-21.1 to 1.4] — P-value and 90% unconditional exact CI was calculated using the model of logit (response) = strata + treatment

4. Primary Outcome: Percentage of Participants Who Achieved Disease Activity Score of 28 Joints Using C-Reactive Protein (DAS28 [CRP]) Response at Day 169
Description: The DAS28 (CRP) was calculated from the number of SJC and TJC using the 28 joints count, The DAS28(CRP) considers 28 of the 68 TJC and 28 of the 66 SJC and participant's global health (GH) using PGA of disease activity using the visual analogue scale (VAS) of 0 (= best), 100 (= worst) plus levels of CRP (milligram/Liter [mg/L]). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) less than (<) 3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Participants with score less than 2.6 were analysed. The percentage of participants were calculated by logistic regression model method.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 29.0 | 17.4
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.108, Logit Response Model; Percent difference = -11.6, 90% CI 2-sided [-23.2 to 0.0] — P-value and 90% unconditional exact CI was calculated using the model of logit (response) = strata + treatment

5. Primary Outcome: Percentage of Participants Who Achieved Health Assessment Questionnaire Disability Index (HAQ-DI) Score Improvement From Baseline and >= 0.25 at Day 169
Description: The HAQ-DI: 20-item scale assessing participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arising, eating, hygiene, walking, reaching, grip, and errands/chores over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range from 0 to 3; where 0 = least difficulty and 3 = extreme difficulty. Participants with change from baseline more than or equal to (>=) 0.25 were reported. The percentage of participants were calculated by logistic regression model method.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 69.0 | 58.7
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.2080, Logit Response Model; Percent difference = -10.3, 90% CI 2-sided [-23.7 to 3.0] — P-value and 90% unconditional exact CI was calculated using the model of logit (response) = strata + treatment

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and Day 169 that were absent before treatment or that worsened relative to pre-treatment state. TEAE and TESAE were reported as per relatedness and severity.
Time Frame: Baseline up to Day 169
Population: The safety population included all participants who received any amount of study medication.
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants
  TEAEs | 29 | 36
  TESAEs | 3 | 2
  Investigational-product-related TEAE | 11 | 12
  Severe TEAE | 3 | 1
  Acute TEAEs | 7 | 5
  Acute Severe TEAE | 1 | 0
  Investigational-product-related TESAE | 2 | 0

7. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Any medically significant change in laboratory evaluations were recorded as adverse events. Following parameters were analyzed for laboratory examination: hematology (leukocytosis, neutropenia, anaemia of chronic disease); serum chemistry (alanine aminotransferase, blood parathyroid hormone, gamma glutamyl transferase, hepatic enzyme, dyslipidaemia, hypercholesterolaemia, hyperglycaemia, hyperlipidaemia, hypertriglyceridaemia); urinalysis.
Time Frame: Baseline up to Day 169
Population: The safety population included all participants who received any amount of investigational product.
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants
  Leukocytosis | 0 | 2
  Neutropenia | 1 | 0
  Anaemia of chronic disease | 1 | 0
  Alanine aminotransferase increased | 2 | 0
  Blood parathyroid hormone increased | 0 | 1
  Gamma-glutamyltransferase increased | 1 | 0
  Hepatic enzyme increased | 2 | 3
  Dyslipidaemia | 2 | 0
  Hypercholesterolaemia | 2 | 0
  Hyperglycaemia | 0 | 1
  Hyperlipidaemia | 0 | 1
  Hypertriglyceridaemia | 0 | 1
  Urinalysis | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included blood pressure, pulse rate, temperature, weight and respiration rate. Vital signs abnormalities reported as TEAEs were reported.
Time Frame: Baseline up to Day 169
Population: The safety population included all participants who received any amount of study medication.
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants
  Hypertension | 0 | 1
  Pyrexia | 2 | 0

9. Secondary Outcome: Number of Participants With Pulmonary Function Test Values Below Threshold Values Based on Percent Change From Baseline at Day 85 and 169
Description: Pulmonary function testing were performed by spirometry to assess forced expiratory volume in 1 second (FEV1), forced expiratory volume in 6 second (FEV6), forced vital capacity (FVC), and diffusing capacity for carbon monoxide (DLCO). FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FEV6 was the maximal volume of air exhaled in the six second of a forced expiration from a position of full inspiration. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. DLCO is a pulmonary function test that measures the partial pressure difference between inspired and expired carbon monoxide. The percentage of predicted values of these pulmonary function tests were calculated based on decreases from baseline and categorized as more than (>) 20% reduction (RD) and absolute value (AV) less than (<) 80% predicted (PR).
Time Frame: Day 85 and 169
Population: The safety population included all participants who received any amount of investigational product. Here "n" signifies participants who were evaluable for this measure for the specified threshold value mentioned parameter for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants
  Day 85: FEV1 > 20% RD (n=64, 63) | 1 | 0
  Day 169: FEV1 > 20% RD (n=64, 64) | 4 | 1
  Day 85: FEV1 > 20% RD and AV < 80% PR (n=64, 63) | 1 | 0
  Day 169: FEV1 > 20% RD and AV < 80% PR (n=64, 64) | 4 | 1
  Day 85: FEV6 > 20% RD (n=54, 55) | 1 | 1
  Day 169: FEV6 > 20% RD (n=54, 56) | 4 | 0
  Day 85: FEV6 > 20% RD and AV < 80% PR (n=54, 55) | 0 | 1
  Day 169: FEV6 > 20% RD and AV < 80% PR (n=54, 56) | 2 | 0
  Day 85: FVC > 20% RD (n=64, 63) | 0 | 0
  Day 169: FVC > 20% RD (n=64, 64) | 2 | 1
  Day 85: FVC > 20% RD and AV < 80% PR (n=64, 63) | 0 | 0
  Day 169: FVC > 20% RD and AV < 80% PR (n=64, 64) | 2 | 1
  Day 85: DLCO > 15-20% RD (n=18, 21) | 1 | 0
  Day 169: DLCO > 15-20% RD (n=22, 23) | 0 | 0
  Day 85: DLCO > 20% RD (n=18, 21) | 1 | 0
  Day 169: DLCO > 20% RD (n=22, 23) | 1 | 0

10. Secondary Outcome: Dyspnea Score at Day 169
Description: Borg dyspnea scale was a validated participant reported outcome assessing participant's perceived difficulty in breathing (dyspnea). The scale ranges from 0 (nothing at all) to 10 (maximal difficulty). Higher scores indicated greater difficulty in breathing.
Time Frame: Day 169
Population: The safety population included all participants who received any amount of investigational product. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 64 | 63
units on a scale | 0.34 (0.81) | 0.42 (0.73)

11. Secondary Outcome: Change From Baseline in Disease Activity Score of 28 Joints Using C-Reactive Protein (DAS28 [CRP]) Score at Day 169
Description: DAS28 (CRP) calculated swollen joint count (SJC) and tender joint count (TJC) using the 28 joints, general health (GH) using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and CRP (milligram per liter [mg/L]). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) less than (<) 3.2 = low disease activity, greater than or equal to (>=) 3.2 to 5.1 = moderate to high disease activity and <2.6= remission.
Time Frame: Baseline and Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
units on a scale
  Baseline (n=68, 70) | 5.72 (0.83) | 5.82 (0.96)
  Day 169 (n=62, 62) | -2.40 (1.42) | -2.11 (1.30)

12. Secondary Outcome: Change From Baseline in Continuous American College of Rheumatology (ACRn) Score at Day 169
Description: ACR score - continuous (ACRn) was defined as the minimum of the percentage improvement in TJC, SJC and the median of the percentage improvements in the other five components of the ACR criteria (participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; disability index of the HAQ; and CRP). Total score range was -100 to 100, where negative numbers indicated worsening and positive numbers indicated improvement. Mean indicates adjusted mean (Adj mean).
Time Frame: Baseline up to Day 169
Population: as for outcome 11
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
units on a scale | 40.49 (5.406) | 33.06 (5.199)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.213, Repeated measures model; Adjusted Mean difference = -7.42, 90% CI 2-sided [-17.24 to 2.40] — An estimate of the treatment difference and its 90% CI was computed by means of repeated measures model, adjusted for baseline and including a treatment by visit interaction term

13. Secondary Outcome: American College of Rheumatology (ACR) Hybrid Score at Day 169
Description: ACR Hybrid score was defined as the minimum of the percentage improvement in TJC, SJC and the median of the percentage improvements in the other five components of the ACR criteria (participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; disability index of the HAQ; and CRP). Total score range was -100 to 100, where negative numbers indicated worsening and positive numbers indicated improvement.
Time Frame: Day 169
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
units on a scale | 49.99 [-9.0 to 98.2] | 41.66 [-1.0 to 90.3]

14. Secondary Outcome: Number of Participants Who Achieved DAS28 (CRP) Response by European League Against Rheumatism (EULAR) Category at Day 169
Description: DAS28 (CRP) response by EULAR category were used to measure individual response as none, moderate, and good, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with baseline DAS28 (CRP) <3.2; moderate response: change from baseline >1.2 with baseline DAS28 (CRP) >=3.2 to less than or equal to (=<) 5.1 or change from baseline >=0.6 to =< 1.2 with baseline DAS28 (CRP) >=3.2 to =<5.1; no response: change from baseline <0.6 or change from baseline >=0.6 and =<1.2 with baseline DAS28 (CRP) >5.1.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants
  No response | 12 | 16
  Moderate response | 28 | 35
  Good response | 28 | 19
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.129, Proportional odds analysis; Odds Ratio (OR) = 0.61, 90% CI 2-sided [0.36 to 1.04] — Odds ratio, 90% CI and p-value were was calculated using proportional odds analysis of response model including treatment as a factor

15. Secondary Outcome: Number of Participants With DAS28 (CRP) Remission and Low Disease Activity at Day 169
Description: DAS28 (CRP) calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and CRP (mg/L). Total score range: 0-9.4, higher score= more disease activity. Remission was defined as less than 2.6 DAS28 (CRP) score. Low disease activity was defined as less than 3.2 DAS28 (CRP) score.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants
  DAS28 (CRP) Remission | 20 | 12
  Low Disease Activity | 28 | 20
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; DAS28 (CRP) remission: p-value estimated from fisher's exact test when number of golimumab or active responders was less than 5; Test type: Superiority or Other; p = 0.108, Regression, Logistic; Percent difference = -11.6, 90% CI [-23.2 to 0.0] — 90% CI was calculated for the treatment difference in proportion of responders using logisitic regression with strata and treatment as factors
Statistical Analysis 2: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; The analysis reported DAS28 (CRP) low disease activity response; Test type: Superiority or Other; p = 0.145, Regression, Logistic; Percent difference = -11.7, 90% CI 2-sided [-24.8 to 1.4] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Time to Onset DAS28 (CRP) Remission at Day 169
Description: The DAS28 (CRP) was calculated from the number of SJC and TJC using the 28 joints count, The DAS28(CRP) considers 28 of the 68 TJC and 28 of the 66 SJC and participant's global health (GH) using PGA of disease activity using the VAS of 0 (= best), 100 (= worst) plus levels of CRP (mg/L). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Participants with score less than 2.6 were analysed. Onset of DAS28(CRP) remission ≤ 2.6 defined as the first study day in which the DAS28 score met the criteria.
Time Frame: Day 169
Population: The mITT population analysis set included all participants who were at risk in the treatment group corresponding to their randomized treatment group. Here, "N" is number of participants analysed for this outcome measure.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 20 | 12
days | 57.0 [29.0 to 112.0] | 113.0 [57.0 to 141.0]
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.328, Log Rank; P-value was calculated using the Log rank test

17. Secondary Outcome: Duration of DAS28 (CRP) Remission at Day 169
Description: The DAS28 (CRP) was calculated from the number of SJC and TJC using the 28 joints count, The DAS28(CRP) considers 28 of the 68 TJC and 28 of the 66 SJC and participant's global health (GH) using PGA of disease activity using the VAS of 0 (= best), 100 (= worst) plus levels of CRP (mg/L). Total score range: 0-9.4, higher score= more disease activity. DAS28 (CRP) <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. Participants with score less than 2.6 were analysed. Duration of DAS28(CRP) remission for each subject was defined as number of days from onset of remission to when the subject was no longer in remission.
Time Frame: Day 169
Population: as for outcome 16
Measure: Mean (Standard Error); unit: days
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 20 | 12
days | 105.0 (0.24) | 69.6 (0.15)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.003, Weibull model; P-value was calculated using an Weibull model

18. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Score of 28 Joints Using Erythrocyte Sedimentation Rate (DAS28 [ESR]) < 2.6 at Day 169
Description: The DAS28 (ESR) calculated SJC and TJC using the 28 joints, GH using participant assessment of disease activity (participant rated arthritis activity using the numerical rating scale with 0 = best, 10 = worst), and the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]). Total score range: 0-9.4, higher score = more disease activity. DAS28 (ESR) <3.2 = low disease activity, >=3.2 to 5.1 = moderate to high disease activity and <2.6= remission. The percentage of participants were calculated by logistic regression model method.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 19.0 | 17.3
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; P-value estimated from fisher's exact test when number of golimumab or active responders was less than 5; Test type: Superiority or Other; p = 0.795, Regression, Logistic; Percent difference = -1.7, 90% CI 2-sided [-12.4 to 9.0] — [estimate comment as in outcome 15, analysis 1]

19. Secondary Outcome: Percentage of Participants Who Achieved Simplified Disease Activity Index (SDAI) Remission at Day 169
Description: The SDAI was the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 - 10 centimetre (cm) VAS; and C-reactive protein (CRP) (milligram per deciliter [mg/dL]). The SDAI total score ranges from 0 to 86, where higher scores indicates greater affection due to disease activity. SDAI remission was defined as a score less than or equal to 3.3. The percentage of participants were calculated by logistic regression model method.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 18.9 | 7.2
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.048, Regression, Logistic; Percent difference = -11.7, 90% CI 2-sided [-21.0 to -2.5] — [estimate comment as in outcome 15, analysis 1]

20. Secondary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Remission at Day 169
Description: The CDAI was the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, patient global assessment and physician global assessment assessed on 0 - 10 cm VAS. The CDAI total score ranges from 0 to 76 where higher scores indicates greater affection due to disease activity. CDAI remission was defined as a score less than or equal to 2.8.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 17.6 | 5.7
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.035, Regression, Logistic; Percent difference = -11.9, 90% CI 2-sided [-20.6 to -3.1] — [estimate comment as in outcome 15, analysis 1]

21. Secondary Outcome: Percentage of Participants With American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Remission at Day 169
Description: The ACR/EULAR remission was defined as swollen joint count (0-66), tender joint count (0-68), CRP (mg/dL) and participant global assessment (0-10) all less than or equal to one.
Time Frame: Day 169
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
percentage of participants | 8.9 | 1.4
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.061, Regression, Logistic; Percent difference = -7.5, 90% CI 2-sided [-13.6 to -1.5] — [estimate comment as in outcome 15, analysis 1]

22. Secondary Outcome: Mean Change From Baseline in Swollen and Tender Joint Count at Day 169
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form, no swelling = 0, swelling =1. Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form, no tenderness = 0, tenderness = 1. Mean here indicates adjusted mean.
Time Frame: Baseline and Day 169
Population: as for outcome 11
Measure: Mean (Standard Error); unit: joint count
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
joint count
  SJC: Baseline (n=68, 70) | 14.49 (0.779) | 14.07 (0.824)
  SJC: Change at Day 169 (n=64, 64) | -10.07 (0.777) | -10.08 (0.747)
  TJC: Baseline (n=68, 70) | 24.93 (1.662) | 25.04 (1.543)
  TJC: Change at Day 169 (n=64, 64) | -15.42 (1.457) | -14.19 (1.399)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in swollen joint count at Day 169; Test type: Superiority or Other; p = 0.993, Repeated measures model; Adjusted mean difference = -0.01, 90% CI 2-sided [-1.33 to 1.32] — An estimate of the treatment difference and its 90% CI was computed by means of repeated measures model, adjusted for baseline and including terms for treatment group, visit and treatment by visit interaction
Statistical Analysis 2: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Analysis reported for change from baseline in Tender joint count at Day 169; Test type: Superiority or Other; p = 0.424, Repeated measures model; Adjusted mean difference = 1.23, 90% CI 2-sided [-1.31 to 3.77] — [estimate comment as in outcome 22, analysis 1]

23. Secondary Outcome: Mean Change From Baseline in Patient Assessment of Pain at Day 169
Description: Participants rated the severity of arthritis pain on a 0 to 100 millimeter (mm) Visual Analogue Scale (VAS), where 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline and Day 169
Population: as for outcome 11
Measure: Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
millimeter (mm)
  Baseline (n=68, 70) | 66.93 (2.352) | 69.81 (2.015)
  Change at Day 169 (n=64, 64) | -29.61 (3.843) | -24.72 (3.727)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.272, Repeated measures model; Adjusted mean difference = 4.89, 90% CI 2-sided [-2.46 to 12.24] — [estimate comment as in outcome 22, analysis 1]

24. Secondary Outcome: Mean Change From Baseline in Patient Global Assessment (PGA) of Disease Activity at Day 169
Description: Participants responded to a question, "Considering all the ways your arthritis affects you, how are you feeling today?" by using a 0 - 100 mm VAS, where 0 = very well and 100 = very poorly.
Time Frame: Baseline and Day 169
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mm
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
mm
  Baseline (n=68, 70) | 67.57 (2.219) | 68.53 (2.212)
  Change at Day 169 (n=64, 64) | -28.50 (3.773) | -24.04 (3.671)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.319, Repeated measures model; Adjusted mean difference = 4.46, 90% CI 2-sided [-2.92 to 11.84] — [estimate comment as in outcome 22, analysis 1]

25. Secondary Outcome: Mean Change From Baseline in Physician Global Assessment of Disease Activity (MDGA) at Day 169
Description: Physician Global Assessment of Arthritis was measured by asking the physician to assess the participant's current arthritis disease activity by placing a vertical line on a 0 to 10 cm VAS, where 0 cm = very good and 10 cm = very bad.
Time Frame: Baseline and Day 169
Population: as for outcome 11
Measure: Mean (Standard Error); unit: centimeter (cm)
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
centimeter (cm)
  Baseline (n=68, 70) | 6.89 (0.159) | 7.04 (0.169)
  Change at Day 169 (n=64, 64) | -4.28 (0.317) | -4.11 (0.307)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.640, Repeated measures model; Adjusted mean difference = 0.16, 90% CI 2-sided [-0.42 to 0.74] — [estimate comment as in outcome 22, analysis 1]

26. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Day 169
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range from 0 to 3; where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Day 169
Population: as for outcome 11
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
units on a scale
  Baseline (n=68, 70) | 1.58 (0.063) | 1.59 (0.070)
  Change at Day 169 (n=64, 64) | -0.59 (0.081) | -0.40 (0.078)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.055, Repeated measures model; Adjusted mean difference = 0.18, 90% CI 2-sided [0.03 to 0.34] — [estimate comment as in outcome 22, analysis 1]

27. Secondary Outcome: Ratio of Change C-Reactive Protein (CRP) at Day 169 to Baseline
Description: The ratio of change from baseline for CRP was analyzed and reported. The CRP is a substance produced by the liver that increases in the presence of inflammation in the body. The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement in underlying disease.
Time Frame: Baseline and Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "N" (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 64 | 64
ratio | 0.5036 (344.0) | 0.5142 (100.9)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.752, Repeated measures model; Adjusted geometric mean ratio = 1.06, 90% CI 2-sided [0.79 to 1.41] — An estimate of the treatment difference and its 90% CI was computed by means of repeated measures model including terms for baseline as a continuous covariate and treatment as a factor was used for the analysis

28. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) at Day 169
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. The farther the red blood cells have descended, the greater the inflammatory response.
Time Frame: Day 169
Population: The mITT population analysis set included all participants in the treatment group corresponding to their randomized treatment group. Here "N" (Number of participants analyzed) signifies those participants who were evaluable for this measure. "n'' signifies participants evaluable for specified category for each arm, respectively.
Measure: Geometric Mean (Standard Deviation); unit: millimeter per hour (mm/h)
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
millimeter per hour (mm/h) | 26.8 (21.0) | 27.8 (20.8)
Statistical Analysis 1: Comparison: Golimumab 50 mg Alternating With Placebo vs Mavrilimumab 100 mg; Test type: Superiority or Other; p = 0.725, Repeated measures model; Adjusted geometric mean ratio = 1.05, 90% CI 2-sided [0.84 to 1.30] — [estimate comment as in outcome 27, analysis 1]

29. Secondary Outcome: Serum Concentrations of Mavrilimumab
Description: Serum concentrations after subcutaneous dose of mavrilimumab were calculated
Time Frame: Baseline, Day 8, 15, 29, 85, 141, and 169
Population: The pharmacokinetic (PK) population included all participants who received mavrilimumab and for whom serum concentrations of mavrilimumab were available for PK data analyses. Here "n" signifies participants who were evaluable for the specified time point for each this arm respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 70
nanogram per milliliter (ng/mL)
  Baseline (n=69) | 0.00 (512.9)
  Day 8 (n=66) | 2837.24 (49.1)
  Day 15 (n=67) | 1084.43 (143.6)
  Day 29 (n=69) | 2094.70 (58.9)
  Day 85 (n=67) | 2886.71 (64.1)
  Day 141 (n=63) | 1731.65 (79.3)
  Day 169 (n=64) | 1701.13 (67.9)

30. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies (ADAs) to Mavrilimumab
Description: Immunogenicity assessment included determination of anti-drug (mavrilimumab) antibodies in serum samples. ADA detection measured by using electrochemiluminescence assays.
Time Frame: Day 1 to Day 169
Population: The immunogenicity population included all participants who received at least 1 dose of mavrilimumab and for whom at least one serum sample for immunogenicity testing was available.
Measure: Number; unit: participants
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Number analyzed (Participants) | 68 | 70
participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Day 169
Description: The safety population included all participants who received any amount of study medication.
Arm/Group | Golimumab 50 mg Alternating With Placebo | Mavrilimumab 100 mg
Serious Adverse Events (participants affected / at risk) | 3/68 | 2/70
Other Adverse Events (participants affected / at risk) | 29/68 | 36/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab 50 mg Alternating With Placebo (N=68) | Mavrilimumab 100 mg (N=70)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab 50 mg Alternating With Placebo (N=68) | Mavrilimumab 100 mg (N=70)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (4) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (2) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (7) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Non-compartmental analyses was not performed for pharmacokinetics parameters due to limited sampling schedule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.